CLINICAL TRIAL: NCT01465893
Title: The Investigation Effect of Vitamin D on Retinal Changes in Patient With Optic Neuritis by Optic Coherence Tomography
Brief Title: Effect of Vitamin D on Retinal Changes in Patient With Optic Neuritis by Optic Coherence Tomography
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Masoud Etemadifar, neurology proffesor, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: isfahan medical university
Record Dates: First submitted 2011-10-28; First posted 2011-11-07 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Optic Neuritis
Keywords: vitamin d
MeSH Terms: conditions — Optic Neuritis | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- vitamin D (Active Comparator): vitamin d 50000/w
  Interventions: Drug: Vitamin D
- control (Sham Comparator): follow up
  Interventions: Drug: Vitamin D withheld

INTERVENTIONS:
Drug: Vitamin D — vitamin D ,50000 unit /week
  Arms: vitamin D
Drug: Vitamin D withheld — do not receive anything
  Arms: control

SUMMARY:
This study examines the effect of vitamin D on Retinal changes in patient with optic Neuritis.

ELIGIBILITY:
Inclusion Criteria:

* age 15-50 years
* no history of demyelinative events
* level of vitamin d below 20 ng/ml
* no pass 10-32 day from starting symptom

Exclusion Criteria:

* using vitamin D supplement

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-07 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
measurement Retinal nerve fiber layer (RNFL) thickness by OCT | 10-32 days after optic neuritis

SECONDARY OUTCOMES:
measurement RNFL thickness by OCT | 6 months after optic neuritis

CONTACTS AND LOCATIONS:
Locations (1):
- Isfahan Medical University, Tehran, Iran

REFERENCES:
- [Derived] Salari M, Janghorbani M, Etemadifar M, Dehghani A, Razmjoo H, Naderian G. Effects of vitamin D on retinal nerve fiber layer in vitamin D deficient patients with optic neuritis: Preliminary findings of a randomized, placebo-controlled trial. J Res Med Sci. 2015 Apr;20(4):372-8. PMID 26109993